CLINICAL TRIAL: NCT03495258
Title: A Prospective Randomized Technology Assessment Trial of Prostate Vaporization Techniques in a Canadian Hospital
Brief Title: Prostate Vaporization Techniques in Canadian Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. J. Curtis Nickel, Professor, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Vaporization
Record Dates: First submitted 2014-06-10; First posted 2018-04-11 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Direct Costs Excluding Capital Equipment Purchase; Operator (Surgeon) Completed Questionnaire; Operative Parameters (Time, Bleeding Etc); Complications (Post-op Retention, Bleeding, Re-admission to Hospital, Infection Etc); 3 Month Efficacy Evaluation (Compared to Baseline) Using Validated Symptom Assessment Tools (See Outcome Metrics for Details)
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clarion Evolve Laser Vaporization System (Experimental): Clarion Evolve Laser Vaporization System
  Interventions: Procedure: Clarion Evolve Laser Vaporization System
- Olympus TURis Plasma Vaporization (Experimental): Olympus TURis Plasma Vaporization
  Interventions: Procedure: Olympus TURis Plasma Vaporization

INTERVENTIONS:
Procedure: Clarion Evolve Laser Vaporization System
  Arms: Clarion Evolve Laser Vaporization System
Procedure: Olympus TURis Plasma Vaporization
  Arms: Olympus TURis Plasma Vaporization

SUMMARY:
Kingston General Hospital is committed to upgrading the surgical treatment platform for benign prostate surgery. Vaporization Surgery, either laser-vaporization or electo-vaporization is becoming a "standard" of therapy for benign prostatic hyperplasia rather than the traditional transurethral resection of the prostate. However many Canadian hospitals have been slow to adopt an updated program because of evolving competing technology systems as well as unknown cost, efficacy, complication and patient/surgeon satisfaction considerations. KGH has been recognized as a centre of excellence in evaluating medical therapy for BPH and studies from the institution have impacted BPH care nationally and abroad. Laser and other state of the art BPH surgical technologies are being purchased by Ontario hospitals, including the local area, with no prospective assessment process. Kingston is uniquely advantaged to undertake a randomized comparative study of two of the most promising technology platforms because the investigators have the experience and expertise to perform the study in a hospital and surgeon naive institution.

The investigators propose to directly compare two vaporization techniques, laser and plasma vaporization systems. The investigators will be able to answer the most important questions in technology introduction and technique into our hospital system - cost, efficacy, safety and satisfaction. The results will inform KGH (and other similar Ontario centres) on the advantage or not (financial and patient care related) of investing in a BPH state of the art vaporization technology.

DETAILED DESCRIPTION:
To comparatively evaluate two state of the art vaporization techniques for transurethral prostatectomy, the Clarion Evolve Laser Vaporization System and the Olympus TURis Plasma Vaporization ("button" electrode) system. Both systems are approved for use by Health Canada for vaporization surgery of the prostate. Both techniques involve a vaporization ablation (laser and plasma mechanism respectively) of the prostate, rather than sequential excision (or cutting) of the prostate performed with our traditional TURP technique. Compared to a TURP, both of the two study techniques involve similar endoscopic access to the prostate, similar anesthetic requirements, similar post-operative catheterization but appear to differ in blood loss (less with vaporization techniques), hospital stay (inpatient stay for TURP compared to outpatient discharge for study techniques) and patient recovery (improved with proposed techniques).

The laser vaporization uses a dual wavelength (980 and 1470 nm) diode laser with a fibre that allows for contact vaporization ablation of the prostate. The hospital already uses a Clarion laser system for urinary stone lithotripsy. Clarion will provide the necessary equipment for this platform for the duration of the trial. The plasma vaporization uses a bipolar high frequency generator for vaporization and coagulation. The procedure is performed using a near-contact hovering technique and the tissue removal process is performed in a similar fashion as TURP. The hospital has recently purchased the Olympus platform and the extra equipment required for this study will be provided by Olympus for the study. These technology systems will be compared in a randomized single blinded controlled study in a "technology naive" hospital with "technology naive" surgeons. The primary outcome will be cost with satisfaction, efficacy, learning curve and safety as key outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male at least 45 years of age.
* Peak urinary flow rate at least 4 ml/sec with a voided volume of at least 125 ml.
* IPPS symptom score ≥ 12 at screening visit.
* Prostate volume on DRE estimated to be > 30cc.
* Voluntarily signed informed consent agreement prior to the performance of any study procedures.

Exclusion Criteria:

* Any prior invasive intervention for BPH.
* PSA level greater than 10 ng/ml at screening without either a negative biopsy or documented explanation of why no biopsy was performed.
* Medical condition unfit for surgery
* History or current evidence of carcinoma of the prostate.
* Documented bacterial prostatitis within the past 3 months.
* Known severe bleeding disorder.
* Unable to follow protocol directions or sign informed consent due to organic brain or psychiatric disease.
* History of alcoholism or any other substance abuse, which, in the opinion of the investigator, would affect compliance with the protocol.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-05; Primary Completion 2016-07-08 (Actual); Study Completion 2016-07-08 (Actual)

PRIMARY OUTCOMES:
Clarion laser vaporization of the prostate | 3 months
  Clarion laser vaporization of the prostate
Olympus plasma vaporization of the prostate | 3 months
  Olympus plasma vaporization of the prostate

CONTACTS AND LOCATIONS:
Overall Officials: Curtis Nickel, MD FRCSC, Principal Investigator — Queen's University
Locations (1):
- Centre for Applied Urological Research, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided